CLINICAL TRIAL: NCT00834730
Title: Comparison of N2O Inhalation and Ketamine IV Injection for Sedation in the Treatment of Laceration of Pediatric Patients.
Brief Title: Comparison of N2O Inhalation and Ketamine in Pediatric PSA
Acronym: PSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N2O
Record Dates: First submitted 2009-02-01; First posted 2009-02-03 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Moderate Sedation; Laceration
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Active Comparator): Ketamine 2mg/kg IV
  Interventions: Drug: N2O gas vs ketamine
- N2O gas (Experimental): 50%-70% N2O gas inhalation
  Interventions: Drug: N2O gas vs ketamine

INTERVENTIONS:
Drug: N2O gas vs ketamine — Ketamine : 2mg/kg IV N2O : 50%-70% N2O gas

SUMMARY:
* Ketamine provides effective and relatively safe sedation analgesia for primary closure of lacerated pediatric patients
* However, deep sedation and adverse effects suggest the opportunity to develop alternative strategies
* We compared the efficacy and adverse effects of ketamine to those of N2O gas for analgesia and anxiolysis during primary repair of lacerated pediatric patients

DETAILED DESCRIPTION:
* There were 32 children who were randomly assigned
* Recovery times were markedly shorter in the N2O group compared with those in the ketamine group (median, 0.0 min (interquartile range [IQR], 0.0-4.0 min) vs. median, 21.5 min (IQR, 12.5-37.5 min), N2O vs. ketamine, respectively, p < 0.05)
* Sedation levels were deeper in the ketamine group than in the N2O group, but pain scales were comparable between groups
* No difference was observed in the satisfaction scores by physicians, parents, or nurses.
* N2O inhalation was preferable to injectable ketamine for pediatric patients because it is safe, allows for a faster recovery, maintains sufficient sedation time, and does not induce unnecessarily deep sedation

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with lacerated wound

Exclusion Criteria:

* Contraindication of ketamine or N2O gas
* A wound around eye and mouth

Ages: 36 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The recovery time (from completion of laceration repair to recovery of mental state) | before discharge

SECONDARY OUTCOMES:
Sedation scale | before discharge
pain scale | before discharge
Side effects | during procedure and bedore discharge and 1day after discharge
Satisfaction of parents and clinicians | before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hee Lee, Professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Lee JH, Kim K, Kim TY, Jo YH, Kim SH, Rhee JE, Heo CY, Eun SC. A randomized comparison of nitrous oxide versus intravenous ketamine for laceration repair in children. Pediatr Emerg Care. 2012 Dec;28(12):1297-301. doi: 10.1097/PEC.0b013e3182768a86. PMID 23187987